CLINICAL TRIAL: NCT00603213
Title: Correlation of Intrathoracic Impedance Measure With Blood Plasma Volume in Congestive Heart Failure
Brief Title: Correlation of Intrathoracic Impedance Measures With Blood Plasma Volume in Congestive Heart Failure
Acronym: Optivol
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Adrian Van Bakel, Professor of Medicine, Medical University of South Carolina
Other Study IDs: HR16840
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Impedance; Optivol Thoracid Fluid Status monitoring system
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 15 mls of blood will be drawn to assay for plasma analytes including but not limited to MMPs, TIMPs and collagen propeptides.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood Volume Analysis, Echocardiogram — Blood Volume Analysis: The use of radioactive tracer to determine plasma volume and red cell mass.
  Echocardiogram is an ultrasound of the heart.
  Other Names: BVA-100, Daxor Corp

SUMMARY:
Congestive heart failure is a condition in which the heart is weakened and is unable to pump enough blood to the organs of the body to meet the demands of the body. At times there may be a buildup of fluid in the lungs, legs or other parts of the body. The accumulation of this fluid has been shown to affect the resistance to flow of the electrical impulses generated in the heart. The purpose of this study is to correlate measurements to the passive flow of electricity generated by the heart within the chest (as measured by the Optivol TFS System) with measurements of the volume of blood in the body.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) affects 5 million people in the United States, with an additional 550,000 cases diagnosed each year. Despite major recent strides in treatment, a diagnosis of CHF still carries significant annual morbidity and mortality. The resultant economic burden associated with the management of this disease has been estimated at $40 billion per year, with 60% - 75% resulting from inpatient management(1). Emergency room visits, frequent outpatient encounters and the hemodynamic monitoring and intensive care associated with inpatient management contribute significantly to this total cost.

Current outpatient heart failure management programs focus on lifestyle changes, pharmacotherapy, and disease awareness, emphasizing self identification of signs and symptoms of volume overload. Despite the best efforts of all involved, frequent unscheduled visits to the outpatient clinic or emergency department remain common, even in those patients participating in formal management programs. Accurate identification of elevated filling pressures and intravascular volume prior to the significant worsening of symptoms remains an elusive goal of management.

Although elevated jugular venous pressure and the presence of a third heart sound have been shown to have prognostic value in patients with heart failure(2), physical exam findings of elevated filling pressures do not reliably correlate with invasive hemodynamics(3).

Invasive measurement of filling pressures and cardiac output with a pulmonary artery catheter has been the gold standard for hemodynamic assessment for decades. However, this method carries significant inherent risks of placement and maintenance and is not well-suited for frequent assessment in the outpatient setting. Development of a method that would accurately and reliably identify hypervolemia and elevated filling pressures prior to the onset of symptoms may allow earlier intervention and have a significant impact on quality of life, morbidity, and mortality in patients with CHF.

Blood volume analysis has been used for over 100 years in the assessment of plasma volume and red cell mass. Earlier techniques relied on dilution of various dyes and were based on the concept that the concentration of a known quantity of dye was inversely proportional to the volume of blood into which it was injected. Later, using the same concept, 51Cr labeled red blood cells and 125I labeled albumen, were developed to measure the red cell and plasma compartments respectively. Although the dual isotope method is considered the gold standard, it is cumbersome and requires at least 6 hours for completion.

A newer, highly automated method using 131I labeled albumen and serial hematocrit measurements (BVA-100, Daxor Corp. New York, NY) has been shown to correlate well with the dual isotope method requiring only 1 ½ hours for completion (Dworkin et al, unpublished data). Additionally, this method can automatically compare measured blood, plasma and red cell volumes to norms based on the sex, weight and height of the patient in the manner of Feldschuh and Enson(4).

Using this method, Androne et al(5) found that 65% of nonedematous CHF patients had unrecognized hypervolemia. More recently, anemia has been shown to be a poor prognostic marker in CHF. In a separate report, Androne et al(6) found that 46% of anemic CHF patients had dilutional anemia vs. 54% with true anemia. The success of targeted therapy may depend on determining whether anemia is dilutional or due to reduced red cell mass. Despite this method's accuracy, it is not practical for the serial measurements required to proactively intervene in a CHF population.

Transthoracic impedance cardiography (ICG) relies on changes in transthoracic electrical impedance when alternating currents are applied across the thorax. Derived measures include stroke volume, cardiac output and thoracic fluid content. Although earlier studies have validated the use of this method in the assessment of intrathoracic volume(7), there have been conflicting results in regard to the correlation of cardiac output (CO) derived from transthoracic ICG and that obtained from more traditional methods such as thermodilution, indicator dye-dilution and the Fick method(8). In addition, the cumbersome nature of serial data acquisition and the realization that derived hemodynamic data may be affected by lead placement make this method less attractive in the ambulatory setting.

Intrathoracic impedance is similar to transthoracic ICG in that it relies on changes in impedance as a surrogate marker of volume status. The technique measures impedance from a right ventricular lead to a pacing/defibrillator case. The technique is not subject to the operator dependent variability of ICG and is well suited to serial measurements in the outpatient setting.

The Optivol® system developed by Medtronic (Minneapolis, MN) employs proprietary software (TFS) that collects and averages impedance values during a specific time period each day to produce the Daily Impedance Value. The TFS software then derives and stores the Daily Mean Impedance, Reference Impedance, and Cumulative Difference from the Daily Impedance Value. The use of predetermined thresholds for the Cumulative Difference from the Daily Impedance Value can provide an early warning of increasing thoracic fluid. This data is accessible to health care practitioners through periodic download in the clinic via interrogation or through Medtronic's web-based CareLink system.

Abraham et al(9) demonstrated that TFS trends are consistent with clinical fluid status in a small group of patients. In addition, a recent study by Yu et al(10) found that intrathoracic impedance is inversely related to pulmonary capillary wedge pressure, and begins to decrease days before the onset of symptoms of CHF.

While data derived from the Optivol® system appears to mirror intrathoracic fluid content, and is useful for determining trends, certain shortcomings remain. First, though changes in intrathoracic impedance may inversely mirror changes in thoracic fluid content, the system provides no absolute reference standard to determine euvolemia in an individual patient. Secondly, it is unclear whether certain concomitant conditions (anemia, COPD) can affect the relationship.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with NYHA II-IV CHF of at least six months duration who have been implanted with a device capable of serial intrathoracic impedance measurement (Optivol®) will be recruited.
* Patients implanted with an Optivol ®device will be eligible for enrollment six months following implantation
* Women of childbearing potential may be included if they have a negative urine pregnancy test at the time of enrollment and agree to use effective contraception throughout the study and for 1 month following their participation

Exclusion Criteria:

* Thoracotomy within previous 3 months
* Chronic pericardial or pleural effusion
* Serum albumen < 2.8 g/dL
* Women who are pregnant or lactating
* Inability or unwillingness to maintain adequate contraception(women of childbearing potential) for the duration of the study and for 1 month following their participation
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with NYHA Class II-IV CHF of at least six months duration who have been implated with a device capable of serial impedance measurement will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
1. correlation between change in intrathoracic impedance and change in total blood volume 2.correlation between change in intrathoracic impedance and change in plasma volume | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VanBakel, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States